CLINICAL TRIAL: NCT01740193
Title: Randomized Prospective Comparison of Analgesic Efficacy of Surgeon Performed IIlioinguinal/Iliohypogastric Blockade With Ultrasound-Guided TAP Blockade in Pediatric Patients Undergoing Unilateral Herniorrhaphy on an Outpatient Basis
Brief Title: Comparison of Two Different Pain Management Techniques in Pediatric Patients Undergoing a Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-1778
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Pain; Inguinal Hernia
Keywords: Pain; Regional Anesthesia; ultrasound; transversus abdominis plane; herniorrhaphy; pediatrics
MeSH Terms: conditions — Pain; Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP Block (Active Comparator)
  Interventions: Procedure: TAP Block
- Ilioinguinal/iliohypogastric blockade (Active Comparator)
  Interventions: Procedure: Ilioinguinal/iliohypogastric blockade

INTERVENTIONS:
Procedure: TAP Block — While the terminal branches of T7 to L1 cannot be visualized under ultrasound as they pass between the internal oblique and the transverse abdominis muscles, they are expected to lie within this plane. The three muscular layers of the abdominal wall, however, can be easily identified under ultrasound guidance. A needle is advanced under ultrasound guidance towards the fascial plane that separates the internal oblique and the transversus abdominis muscles, at which point local anesthetic is deposited under direct visualization.
  Other Names: transversus abdominis plane block
  Arms: TAP Block
Procedure: Ilioinguinal/iliohypogastric blockade — Ilioinguinal and iliohypogastric blockade is performed as an injection after palpation of the anterior superior iliac spine followed be a perceived loss of resistance with insertion of the needle, or may be infiltrated locally following herniorrhaphy exposure as anatomic landmarks can prove to be difficult to locate in the anesthetized pediatric patient.
  Arms: Ilioinguinal/iliohypogastric blockade

SUMMARY:
The purpose of this research study is to find the best way to decrease pain in children right after surgery whom have had their hernia fixed. Right now, there are two different ways surgeons and anesthesia providers try to decrease pain. It is not clear if one way is better than the other. The method used is often chosen by which one the doctor has more experience using. The Investigator plans to find out if one of the methods is more effective and/or safer than the other method.

The results of this study will help learn how to best control pain in children having surgery for hernia repair.

DETAILED DESCRIPTION:
Unilateral inguinal herniorrhaphy is a commonly performed surgical procedure in the pediatric population. Multimodal anesthesia consisting of systemic narcotics, surgical wound infiltration with local anesthetic and ilioinguinal and/or iliohypogastric nerve blockade has traditionally been employed to achieve acceptable analgesia. Recently, ultrasound-based studies have demonstrated that blind abdominal wall injections are done with poor accuracy. Ultrasound-guided alternatives, such as the transverses abdominis plane (TAP) block, may improve analgesic efficacy and patient comfort in the post-operative period when compared to blind landmark based nerve blockade. There has been increasing utilization of the TAP block in the adult population due to the described ability to provide effective blockade of the thoracolumbar spinal nerves innervating the abdominal wall. We propose a randomized prospective evaluation of the analgesic efficacy comparing surgeon performed ilioinguinal/iliohypogastric block with ultrasound-guided TAP blockade in healthy ASA I and II pediatric patients undergoing unilateral herniorrhaphy on an outpatient basis.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female;
* The subject is of any racial and ethnic groups;
* The subject is age 12 months to 10 years (inclusive);
* The subject weighs more than 8.0 kg (inclusive of the eighth kilogram);
* The subject is scheduled for the following: Unilateral herniorrhaphy scheduled on an out-patient basis, and not being performed in conjunction with any other surgical procedures;
* The subject is American Society of Anesthesiologists (ASA) patient classification I-II
* The subject's legally authorized representative has given written informed consent to participate in the study and when appropriate, the subject has given assent or consent to participate.

Exclusion Criteria:

* Additional surgical procedures are being performed concurrently;
* The subject is ASA classification > II;
* The subject has pre-existing allergies to local anesthetics;
* The subject receives midazolam as a premedication;
* The subject has an imminent life threatening condition that impacts the ability to obtain informed consent;
* The subject has any other condition, which in the opinion of the principal investigator, would not be suitable for participation in the study.

Ages: 12 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2012-08; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Efficacy Outcome | Participants will be followed for the duration of post-anesthesia care unit stay, an expected average of 2 hours
  Worst FLACC score observed in the post-anesthesia care unit by the research coordinator during the first post-operative hour

SECONDARY OUTCOMES:
Efficacy Outcome - Length of Recovery Room | participants will be followed for the length of the surgical procedure, an expected average of 1.5 hours
  time required for the patient to meet discharge criteria
Confounding Variable - Electrocautery | participants will be followed for the length of the surgical procedure, an expected average of 1.5 hours
  whether or not cautery was used as a measure of surgical technique
Confounding Variable - Surgical dissection | participants will be followed for the length of the surgical procedure, an expected average of 1.5 hours
  length of surgical procedure as an indicator of the extent of surgical dissection performed
Confounding Variable - Length of time for TAP | participants will be followed for the length of the surgical procedure, an expected average of 1.5 hours
  length of time required to perform TAP block
Efficacy Outcome - Post-operative Calls | participants will be followed for 48 hours after procedure
  Phone calls made to surgeons regarding parental concern of post-operative pain forty-eight hours post-operatively
Outcome Measure - Number of patients with post-operative complications | participants will be followed for 48 hours after procedure
  presence of post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Furstein, CRNA, DNAP, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hosptial Medical Center - Liberty Campus, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Niraj G, Searle A, Mathews M, Misra V, Baban M, Kiani S, Wong M. Analgesic efficacy of ultrasound-guided transversus abdominis plane block in patients undergoing open appendicectomy. Br J Anaesth. 2009 Oct;103(4):601-5. doi: 10.1093/bja/aep175. Epub 2009 Jun 26. PMID 19561014
- [Background] Fredrickson M, Seal P, Houghton J. Early experience with the transversus abdominis plane block in children. Paediatr Anaesth. 2008 Sep;18(9):891-2. doi: 10.1111/j.1460-9592.2008.02591.x. No abstract available. PMID 18768050
- [Background] Aveline C, Le Hetet H, Le Roux A, Vautier P, Cognet F, Vinet E, Tison C, Bonnet F. Comparison between ultrasound-guided transversus abdominis plane and conventional ilioinguinal/iliohypogastric nerve blocks for day-case open inguinal hernia repair. Br J Anaesth. 2011 Mar;106(3):380-6. doi: 10.1093/bja/aeq363. Epub 2010 Dec 21. PMID 21177284
- [Background] Fredrickson MJ, Seal P. Ultrasound-guided transversus abdominis plane block for neonatal abdominal surgery. Anaesth Intensive Care. 2009 May;37(3):469-72. doi: 10.1177/0310057X0903700303. PMID 19499870
- [Background] Groudine SB, Fisher HA, Kaufman RP Jr, Patel MK, Wilkins LJ, Mehta SA, Lumb PD. Intravenous lidocaine speeds the return of bowel function, decreases postoperative pain, and shortens hospital stay in patients undergoing radical retropubic prostatectomy. Anesth Analg. 1998 Feb;86(2):235-9. doi: 10.1097/00000539-199802000-00003. PMID 9459225
- [Background] Hadzic A, New York School of Regional Anesthesia.: Textbook of regional anesthesia and acute pain management. New York: McGraw-Hill, Medical Pub. Division; 2007.